CLINICAL TRIAL: NCT06011265
Title: Does Mirabegron Increase the Body Heat Generated by the Nervous System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Christopher Bell (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2981
Record Dates: First submitted 2023-07-24; First posted 2023-08-25 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Thermoregulation
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Crossover with a washout of at least 10 days
Who Masked: Participant
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirabegron + Isoproterenol (Experimental): 100mg oral + Isoproterenol IV Infusion; 3 doses, 6, 12, 24ng/ kg Fat Free Mass
  Interventions: Drug: Myrbetriq 25Mg Extended-Release Tablet
- Placebo + Isoproterenol (Placebo Comparator): Empty Capsule + Isoproterenol IV Infusion; 3 doses, 6, 12, 24ng/ kg Fat Free Mass
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Myrbetriq 25Mg Extended-Release Tablet — Participants take 4x 25mg Myrbetriq 25Mg Extended-Release Tablet orally.
  Arms: Mirabegron + Isoproterenol
Drug: Placebo — Participants take empty capsule orally
  Arms: Placebo + Isoproterenol

SUMMARY:
Acute mirabegron administration has been shown to increase brown fat activity in humans. Long-term mirabegron administration upregulates brown fat, and appears to improve glucose regulation, and change skeletal muscle phenotype.

DETAILED DESCRIPTION:
The Undersea Medicine Program at the Office of Naval Research has invited Indiana University, Rutgers and Colorado State University, to explore the potential of the medication, Mirabegron, to improve the cold tolerance of Navy personnel. Indiana University will submit the formal application for research funding. Research activities at Colorado State University will be supported by a sub-contact from Indiana University.

The project will address four hypotheses. One of these hypotheses will be investigated exclusively at Colorado State University during the second year of the project. The proposed activities at Colorado State University will be unique; the link to activities performed by Indiana University and Rutgers is thematic only.

Specialized Navy personnel are required to undertake duties while immersed in cold water for prolonged periods. These dives regularly require the use of external thermal protection (i.e., wet suits and dry suits). However, external thermal protection during prolonged cold-water diving is often times insufficient to maintain body temperature and thermal comfort, thereby potentially negatively impacting the safety and success of diving missions. Accordingly, developing an alternative strategy that can improve tolerance to cold-water immersion is of important interest to Navy divers and special forces. In this regard, the pharmaceutical, mirabegron, may hold considerable promise to mitigate the negative effects of cold-water immersion on cold-water tolerance by increasing thermogenesis (the generation of heat). Mirabegron (Myrbetriq®, extended-release tablet, Astellas Pharma), is a medication approved by the Food and Drug Administration for the treatment of overactive bladder. In 2020, it was the 160th most commonly prescribed medication in the United States, with more than three million prescriptions. The mechanism of action is stimulation of beta-3-adrenergic receptors (receptors that are usually stimulated by the sympathetic nervous system). Mirabegron is also known to stimulate brown fat, a metabolically active, heat-generating tissue. The overall goals of the project are to determine the efficacy of acute mirabegron administration to improve cold tolerance and determine if mirabegron can accentuate thermogenesis during sympathetic activation.

ELIGIBILITY:
Inclusion Criteria:

* age 18-40 years,
* regular participation in more than 150 minutes of moderate intensity exercise, every week, during the previous two years.

Exclusion Criteria:

* History of autonomic, cardio-pulmonary, and/or metabolic disease (including heart failure, hypertension, arrhythmia, vascular disease, and/or diabetes)
* contraindication for mirabegron ingestion, such as previously diagnosed liver and/or kidney dysfunction,
* use of medication that may unfavorably interact with mirabegron, including thioridazine (Mellaril™ and Mellaril-S™), flecainide (Tambocor®), propafenone (Rythmol®), digoxin (Lanoxin®) and solifenacin succinate (VESIcare®)
* pregnancy or breast feeding
* habitual use of tobacco/nicotine products (2 or more uses within the previous month)
* any type of bladder dysfunction, taking medication related to bladder issues, or a history of bladder issues.
* Sulfite Allergy '

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in metabolic rate compared to baseline during each stage as measured by indirect calorimetry | Immediately after each infusion
  Participants will undergo a 45 minute resting metabolic rate assessment and then consume Mirabegron or Placebo. Afterwards, they will undergo three 30 minute infusions of Isoproterenol consisting of doses of 6, 12, and 24ng/kg FFM
Change in temperature among the top 10% of hottest pixels as identified via thermal camera and FLIR research software in the supraclavicular region during each isoproterenol infusion. | Immediately after each infusion.
  At the conclusion of each of the 3 isoproterenol infusions, participants will have thermal images taken of their supraclavicular region to identify brown fat activation.
Change in core temperature measured via oral thermometer during each stage. | Immediately after each infusion.
  Core temperature will be measured via oral thermometer at the conclusion of each of the three isoproterenol infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bell, Ph.D., Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No